CLINICAL TRIAL: NCT00320112
Title: Improving Insulin Therapy With Enhanced Care Management and Peer Support
Brief Title: Improving Insulin Therapy With Enhanced Care Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IIR 04-239
Record Dates: First submitted 2006-04-27; First posted 2006-05-03 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes
Keywords: telemedicine; case management; insulin; self-care
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reciprocal Diabetes Peer Support program (Experimental): peers are paired during the group visit and are encouraged to speak with their partner at least once a week for the 6 month duration of the study.
  Interventions: Behavioral: Reciprocal Diabetes Peer Support Program; Behavioral: group outpatient counseling visits
- Nurse Case Management (Other): patients are not paired in the NCM arm. they are provided with educational session on diabetes management and informed of case management services.
  Interventions: Behavioral: Nurse Case management

INTERVENTIONS:
Behavioral: Reciprocal Diabetes Peer Support Program — participants are paired with another age-matched participation. Paired peer partners were encouraged to talk weekly using a telephone platform that recorded call frequency and duration and provided automated reminders promoting peer contact.
  Arms: Reciprocal Diabetes Peer Support program
Behavioral: Nurse Case management — patients are not paired in the NCM arm attended a 1.5 hour session to receive education on care manager services and diabetes educational materials and be assigned to a nurse care manager with whom they were encouraged to follow-up regularly.
  Arms: Nurse Case Management
Behavioral: group outpatient counseling visits — Participants in the peer group were also offered three optional 1.5 hour patient-driven group sessions at month 1, 3, and 6
  Arms: Reciprocal Diabetes Peer Support program

SUMMARY:
VA diabetes patients often have difficulty managing their self-care and accessing clinic-based services; many also lack social support to help them meet the demands of their illness. Enhanced support is especially important when undertaking and sustaining new challenging self-care tasks, such as initiating or intensifying insulin treatment regimens. Although some VAs have implemented telephone nurse care management programs supported by automated calling services, many are reluctant to adopt these models due to nursing shortages.

DETAILED DESCRIPTION:
Background:

VA diabetes patients often have difficulty managing their self-care and accessing clinic-based services; many also lack social support to help them meet the demands of their illness. Enhanced support is especially important when undertaking and sustaining new challenging self-care tasks, such as initiating or intensifying insulin treatment regimens. Although some VAs have implemented telephone nurse care management programs supported by automated calling services, many are reluctant to adopt these models due to nursing shortages.

Objectives:

This randomized trial will evaluate an intervention using a low-cost interactive voice response (IVR) exchange system to promote peer-to-peer communication among diabetes patients initiating or increasing insulin therapy under medical guidance. The intervention is based on research demonstrating the positive impact of peer support on chronic disease outcomes and self-care behaviors, our own prior studies demonstrating the effectiveness of IVR-based self-management supports for VA diabetes patients, and a successful pilot study demonstrating VA diabetes patients' willingness to participate in IVR-facilitated peer support. The Specific Aims are: (1) To evaluate the effect of IVR-facilitated peer support on diabetes patients' glycemic control (including their A1c levels, insulin doses, hypo- and hyperglycemic symptoms) and use of VA care; (2) To assess the impact of IVR-facilitated peer support on patient-centered outcomes, including patients' satisfaction with care, perceived social support, diabetes-specific quality of life, and self-care behaviors; and (3) To identify patient characteristics associated with participation and use of IVR peer support, and mediators of the intervention's impact on patient outcomes.

Methods:

324 diabetes patients with inadequate glycemic control who are candidates for insulin initiation or intensification will be recruited from 2 VA facilities (Ann Arbor, and Toledo). We will pair eligible patients based on age, gender, and whether they are initiating or increasing insulin. Pairs will be randomized to either: 1) usual care; or 2) usual care in conjunction with the IVR-based peer support program. After their orientation, intervention participants will be asked to communicate weekly with their partner using the IVR exchange. The IVR service is designed to allow patients to communicate without divulging their home phone number, experiencing toll charges, or being responsible for insuring that contacts occur without the assistance of reminder prompts. Intervention patients who have achieved adequate glycemic control at their 6-month follow up will be encouraged to select a new treatment goal. Patients will continue to participate in weekly IVR calls for 6 months. Research staff will monitor the process via the Internet, and outcomes will be measured at six months. The primary endpoint will be HbA1c levels at 6 and 12-months. Secondary endpoints include other physiological measures and patient-centered outcomes. The intervention is designed to interact with standard outpatient VA staffing models. We will develop detailed training materials that facilitate implementation in other facilities and work with clinical managers to facilitate roll-out if the intervention is found to be effective.

Status:

Recruitment of participants is complete as well as most preliminary data analyses. 12 month data is now being analyzed.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* HbA1c > 7%
* age > 21

Exclusion Criteria:

* substance abuse disorder
* serious psychiatric illness
* serious hearing loss
* life expectancy < 12 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2007-02; Primary Completion 2009-10 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Piette, PhD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Heisler M, Vijan S, Makki F, Piette JD. Diabetes control with reciprocal peer support versus nurse care management: a randomized trial. Ann Intern Med. 2010 Oct 19;153(8):507-15. doi: 10.7326/0003-4819-153-8-201010190-00007. PMID 20956707

RESULTS

PARTICIPANT FLOW:
Groups:
- Reciprocal Diabetes Peer Support Program (RPS): participants in the intervention arm are paired with a peer
  Peer-support telephone calls: peers are paired during the group visit and are encouraged to speak with their partner at least once a week for the 6 month duration of the study.
  group outpatient counseling visits: participants are given the option to attend 3 optional group visits with other participants and case managers. this gives them the opportunity to ask any diabetes related questions of nurses or other participants who have diabetes.
- Nurse Case Management: participants were randomized to receive usual care with an initial educational session to review lab results and discuss any questions related to educational handouts. particpants were also provided information about nurse case managements services and encouraged to use the service regularly.
Period: Overall Study
Arm/Group | Reciprocal Diabetes Peer Support Program (RPS) | Nurse Case Management
Started | 125 | 119
Completed | 117 | 114
Not Completed | 8 | 5
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Population: 125 participants were randomized to Reciprocal Peer Support (RPS), and 119 to Nurse case management (NCM).
Groups:
- Receiprocal Peer Support: participants in the intervention arm are paired with a peer
  Peer-support telephone calls: peers are paired during the group visit and are encouraged to speak with their partner at least once a week for the 6 month duration of the study.
  group outpatient counseling visits: participants are given the option to attend 3 optional group visits with other participants and case managers. this gives them the opportunity to ask any diabetes related questions of nurses or other participants who have diabetes.
- Nurse Case Management: participants were randomized to receive usual care with an initial educational session to review lab results and discuss any questions related to educational handouts
- Total: Total of all reporting groups
Arm/Group | Receiprocal Peer Support | Nurse Case Management | Total
Number analyzed (Participants) | 125 | 119 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (6.1) | 62.3 (6.6) | 62.0 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 125 | 119 | 244
Race/Ethnicity, Customized [Number; unit: participants]
  White, non-Hispanic | 99 | 98 | 197
  Hispanic | 5 | 2 | 7
  African American | 11 | 11 | 22
  Other | 9 | 5 | 14
  unkwown | 1 | 3 | 4
Education [Number; unit: participants]
  Some High School, High School | 34 | 35 | 69
  at least some college, technical\vocational school | 91 | 83 | 174
  unknown | 0 | 1 | 1
Annual Income [Number; unit: participants]
  less than or equal to $30,000 | 78 | 71 | 149
  greater than or equal to $31,000 | 46 | 41 | 87
  other or unknown | 1 | 7 | 8
Social Support [Number; unit: participants]
  Lives with a spouse | 82 | 84 | 166
  Lives alone | 29 | 22 | 51
  Other | 14 | 13 | 27
Anti-hyperglycemic Medications [Number; unit: participants]
  Only oral diabetes medication | 55 | 53 | 108
  Insulin, + or - oral medication | 70 | 66 | 136
Self-Rated General Health Status - Fair or Poor Health [Number; unit: participants] | 59 | 64 | 123
HbA1c [Mean (Standard Deviation); unit: percent HbA1c] | 8.02 (1.32) | 7.93 (1.40) | 7.98 (1.40)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 140.3 (18.6) | 136.4 (16.9) | 138.4 (17.9)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 77.1 (11.5) | 75.8 (10.7) | 76.5 (11.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycemic Control (HbA1c)
Description: The primary outcome was change between baseline and six-month Hemoglobin A1c (HbA1c), measured with a Bayer DCA 2000+ point-of-care analyzer.
Time Frame: 6 months (baseline to 6 months)
Population: Peer Support group: 117 of the 125 provided 6 month data and 113 provided physiologic measures. Nurse Case management participants: 114 of 119 provided 6 month data and 103 provided follow-up physiologic measures.
Measure: Mean (Standard Deviation); unit: percent HbA1c
Groups:
- Reciprocal Peer Support Group: participants in the intervention arm are paired with a peer
  Peer-support telephone calls: peers are paired during the group visit and are encouraged to speak with their partner at least once a week for the 6 month duration of the study.
  group outpatient counseling visits: participants are given the option to attend 3 optional group visits with other participants and case managers. this gives them the opportunity to ask any diabetes related questions of nurses or other participants who have diabetes.
- Nurse Case Management Group: Nurse Case Management group was offered an educational session with nurse case managers on diabetes and informed of case management services. they were encouraged to utilize this service regularly.
Arm/Group | Reciprocal Peer Support Group | Nurse Case Management Group
Number analyzed (Participants) | 113 | 103
percent HbA1c
  Baseline percent A1c | 8.02 (1.32) | 7.93 (1.40)
  6 month percent A1c | 7.73 (1.32) | 8.22 (1.74)
Statistical Analysis 1: Comparison: Reciprocal Peer Support Group vs Nurse Case Management Group; Test type: Superiority or Other; p = 0.004, Regression, Linear — no differences between arms in baseline characteristics at <0.1 level, further analyses adjusted for variables that could influence the outcome like insulin use, age, commodities. because no differences in results, unadjusted analyses are reported; we used STATA 11's xtmixed command, which fits multi-level mixed-effects linear regression models, with clustering by assigned pairs; Mean Difference (Final Values) = -0.58

2. Secondary Outcome: Change in Systolic Blood Pressure Measure
Description: secondary outcome measure was change in blood pressure comparison of peer support group and nurse case management group from baseline to six months
Time Frame: change in blood pressure at 6 months
Population: comparison of blood pressure measure taken at baseline and then again at 6 months among the two groups. as noted, 113 peer support participants provided physiologic measures at 6 months and 103 of 119 from the nurse management group provided physiologic measures at 6 months.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Change in Systolic BP at 6 Months for Peer Support Group: change in systolic blood pressure from baseline to six months among participants in the peer support group
- Change in Systsolic at 6 Months for Nurse Mgt Group: change in systolic blood pressure from baseline to six months in the nurse case management group
Arm/Group | Change in Systolic BP at 6 Months for Peer Support Group | Change in Systsolic at 6 Months for Nurse Mgt Group
Number analyzed (Participants) | 113 | 103
mmHg
  baseline systolic blood pressure | 140.3 (18.6) | 136.4 (16.9)
  6 month systolic blood pressure | 136.9 (16.8) | 135.0 (17.7)
Statistical Analysis 1: Comparison: Change in Systolic BP at 6 Months for Peer Support Group vs Change in Systsolic at 6 Months for Nurse Mgt Group; Test type: Superiority or Other; p = .91, Regression, Linear — this is a priori design

3. Secondary Outcome: Change in Diastolic Blood Pressure
Description: change in diastolic blood pressure was measured at 6 months
Time Frame: 6 months from baseline
Population: As noted earlier, for physiologic measures only 113 of the 125 peer support participants were able to provide 6 month follow-up data and 103 of 119 nurse management group provided 6 month follow-up data.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Reciprocal Peer Support Group: participants are age-matched with a peer and asked to talk with each other weekly using a telephone support sytem
- Nurse Case Management Group: participants in the nurse case management group receive initial educational session on diabetes and information bout case management services. they are encouraged to contact their nurse case manager regularly.
Arm/Group | Reciprocal Peer Support Group | Nurse Case Management Group
Number analyzed (Participants) | 113 | 103
mmHg
  baseline diastolic blood pressure | 77.1 (11.5) | 75.8 (10.7)
  6 month diastolic blood pressure | 76.8 (11.9) | 76.1 (10.6)
Statistical Analysis 1: Comparison: Reciprocal Peer Support Group vs Nurse Case Management Group; Test type: Superiority or Other; p = 0.10, Regression, Linear

4. Secondary Outcome: Number of Participants With Insulin Starts at 6 Months
Description: the number of insulin starts at 6 months from baseline.
Time Frame: 6 months (baseline to 6 months follow-up)
Population: medical charts were reviewed to obtain this information and all participant charts were reviewed
Measure: Number; unit: participants
Groups:
- Reciprocal Peer Support Group: patients were age-matched and assigned to a peer. they were asked to make weekly calls using a telephone support system to check in and discuss their diabetes
- Nurse Case Management Grouop: patients were provided an educational session and discussed nurse case management services. participants were encouraged to meet wit their case manager regularly.
Arm/Group | Reciprocal Peer Support Group | Nurse Case Management Grouop
Number analyzed (Participants) | 125 | 119
participants | 8 | 1
Statistical Analysis 1: Comparison: Reciprocal Peer Support Group vs Nurse Case Management Grouop; Test type: Superiority or Other; p = 0.02, Regression, Linear

ADVERSE EVENTS:
Time Frame: adverse event information was collected through-out the course of a participants enrollment in the study - 6 months
Groups:
- Reciprocal Peer Support Intervention: participants in the intervention arm are paired with a peer
  Peer-support telephone calls: peers are paired during the group visit and are encouraged to speak with their partner at least once a week for the 6 month duration of the study.
  group outpatient counseling visits: participants are given the option to attend 3 optional group visits with other participants and case managers. this gives them the opportunity to ask any diabetes related questions of nurses or other participants who have diabetes.
- Nurse Case Management Intervention: participants were randomized to receive usual care with an initial educational session to review lab results and discuss any questions related to educational handouts
Arm/Group | Reciprocal Peer Support Intervention | Nurse Case Management Intervention
Serious Adverse Events (participants affected / at risk) | 2/125 | 1/119
Other Adverse Events (participants affected / at risk) | 0/125 | 0/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reciprocal Peer Support Intervention (N=125) | Nurse Case Management Intervention (N=119)
Death (General disorders) | 2 (2) | 1 (1) — Cause of death was unknown to study team

LIMITATIONS AND CAVEATS:
1. study only included male patients.
2. intervention only lasted six months.
3. the nature of the intervention prevented blinding to treatment group.
4. A final limitation is the relatively low rate of uptake of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No